CLINICAL TRIAL: NCT06589050
Title: The Effects of Two Foot Strengthening Interventions on Toe Flexor Strength and Jumping Performance in Vocational Ballet Dancers: A Randomized Controlled Trial
Brief Title: Improving Foot Strength in Vocational Ballet Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Elmhurst Ballet School, Birmingham (Unknown); German Sport University, Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5/24/AS/UOW
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Toe Flexor Strength
Keywords: Toe flexor strength; Foot; Dance; Jumping performance

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled study. Participants will be randomly assigned to one of three parallel groups (two experimental groups and one control group) with a 1:1:1 ratio. To balance the covariates of age and sex among the three groups, a computer-based program will perform stratified randomization within three blocks.
Masking Description: After the participants have completed the pre-measurements, they will be assigned to their group allocation. The intervention´s nature precludes blinding the participants and the trainer; however, a supervisor will monitor data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Toe flexor device" experimental group (Experimental): Participants will complete:
  * 3 sets of 15 repetitions with a 90-second break between each set.
  * Tempo 2-0-2-0
  * 4 times per week
  * Progression will be achieved by increasing the stiffness of the elastic band whenever the participant can perform 15 repetitions without great effort.
  Interventions: Other: "Toe flexor device" experimental group
- "Inclined Heel Rise" experimental group (Experimental): Participants will complete:
  * 3 sets of 10 to 15 repetitions with a 90-second break between each set.
  * Tempo 2-0-2-0
  * 4 times per week
  * Progression will be achieved by increasing the number of repetitions to 15 and then adding weights to be held in the ipsilateral hand.
  Interventions: Other: "Inclined Heel Rise" experimental group
- Control group (No Intervention): The control group will continue with the ballet school's normal training schedule.

INTERVENTIONS:
Other: "Toe flexor device" experimental group — This intervention group will perform toe flexion using a toe flexor (TF) device, which facilitates the shortening and stretching of the TF muscle-tendon units (MTUs) against resistance bands. While seated, participants will push a pedal down with their toes over two counts and release it over two counts.
  Arms: "Toe flexor device" experimental group
Other: "Inclined Heel Rise" experimental group — This intervention group will perform single-leg heel rises on an inclined platform. Participants will place their hands against a barre for balance support, lift their heels over two counts, and lower them over two counts.
  Arms: "Inclined Heel Rise" experimental group

SUMMARY:
Professional dancers subject their feet to high forces through frequent jumping, repeated heel rises, insufficient shoe cushioning, and a high degree of foot mobility. To prevent injuries and improve jumping performance, dancers are recommended to strengthen the muscles of the lower extremities.

The foot muscles, especially the toe flexors, play an important role as shock absorbers and motors for the foot by absorbing and generating mechanical energy, which is essential for human locomotion. Furthermore, they serve as a link between the powerful leg extensor muscles and the ground, transmitting the energy generated by the larger muscle groups. This makes them essential components of overall athletic performance. However, the impact of foot muscle strength on dancers´ jumping performance remains uncertain. Therefore, the aim of this study is to investigate the effectiveness of two training programs designed to strengthen the toe flexor muscles in dancers. For this project, a 6.5-week intervention with ballet students from a vocational ballet school is planned. Before and after the intervention, all study participants will perform tests to assess foot muscle strength and jumping performance.

DETAILED DESCRIPTION:
This study aims to develop two different toe flexor (TF) exercise programs for vocational dancers to enhance TF strength and jumping performance. It is hypothesized that i) both training programs increase TF strength and jumping performance, ii) horizontal jumps are more affected than vertical jumps, and iii) the TF exercise program with the TF strengthening device has a greater impact on TF strength.

Participants

Participants will be recruited from a vocational ballet school via an email detailing the study outline. They and their legal guardians (for participants under 18 years old) will be informed of the potential risks and benefits of the study. They will provide written informed consent prior to the measurements. Participants will then be assigned to either a control group, a toe flexor device experimental group, or a heel rise experimental group. The schedule includes three and a half weeks of training, a 12-day break due to the school schedule, followed by another three weeks of training. This will result in a total of 26 training sessions. An experienced trainer will supervise all training sessions. The control group will continue with the ballet school´s normal training schedule.

Data collection and management

An intervention protocol will be kept to collect information on compliance and progression of the training, such as the number of repetitions and the resistance applied. Data analysis will be performed according to the intention-to-treat (ITT) principle, in which participants are analyzed according to their original treatment group assignment. An additional researcher will manage reporting for adverse effects (such as delayed onset muscle soreness) and adverse events. All data collected in this study will be anonymized, personal identifiers removed, and data coded to protect the identities of the participants.

Sample size

Due to the study´s novel character, no sample size calculations have been conducted. To the researchers' best knowledge, no comparable protocols to improve TF strength have been investigated, so a sample size calculation was not warranted. The study is, therefore, exploratory.

Statistical analysis

Variables will be presented as the mean ± standard deviation. The Shapiro-Wilk test will be performed to assess the normality of the measured variables. Repeated-measures Analysis of Variance (ANOVA) with Bonferroni correction will be used to analyze variables across different times and groups. Non-normally distributed variables will be analyzed using Friedman ANOVA and Kruskal-Wallis ANOVA, with multiple comparisons of mean ranks for individual comparisons. Statistical analyses will be performed using IBM SPSS Statistics for Windows (Version 29.0), and the statistical significance level will be set to .05. If the primary and/or secondary outcomes yield null findings, equivalence testing will be conducted to determine whether the intervention is equivalent to the usual training (control group). The two one-sided tests (TOST) procedure will be applied, using either standardized differences (e.g., Cohen's d) or raw differences.

ELIGIBILITY:
Inclusion Criteria

* Being a ballet student at the Elmhurst Ballet School.
* Aged 14 to 19.
* Written informed consent (by the participant and/or their legal guardian).

Exclusion Criteria:

* Any recent lower leg or foot injuries.
* Chronic pain in the lower extremities.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary isometric contraction (MVIC) of the toe flexors muscles | Measurements will be performed one week prior to and one week after the intervention.
  The post-intervention difference between the three groups in MVIC of the toe flexors measured with a custom-made toe flexor dynamometer in a seated position (90° angle in the hips and knees) where the foot is secured with a strap. Participants will push with their toes against a pedal and hold this isometric contraction for 2-3 seconds. The strength will be normalized by body weight (N/kg).

SECONDARY OUTCOMES:
Vertical jump - Countermovement jump (CMJ) - Jump height (cm) | Measurements will be performed one week prior to and one week after the intervention.
  Participants will perform three CMJs on a Hawkin Dynamics force plate. They will stand upright on the plate and be instructed to jump as high as possible with their hands positioned on their hips.
Vertical jump - CMJ - changes in force parameters | Measurements will be performed one week prior to and one week after the intervention.
  Participants will perform three CMJs on a Hawkin Dynamics force plate. The variables collected will be peak power (W), peak propulsive force (N), and peak landing force (N).
Vertical jump - Sauté jump - jump height (cm) | Measurement will be performed one week prior to and one week after the intervention.
  Participants will perform three sautés on a Hawkin Dynamics force plate. They will perform a ballet-specific jump in an upright position with the legs externally rotated. Participants will be instructed to jump as high as possible.
Vertical jump - Sauté - changes in force parameters | Measurements will be performed one week prior to and one week after the intervention.
  Participants will perform three sautés on a Hawkin Dynamics force plate. The variables collected will be peak power (W), peak propulsive force (N), and peak landing force (N).
Horizontal jump - Long jump - jump distance (cm) | Measurements will be performed one week prior to and one week after the intervention.
  Participants will perform three horizontal long jumps with their hands positioned on their hips. The distance of the jumps will be measured (cm).

OTHER OUTCOMES:
End User Questionnaire | After the intervention, up to one hour.
  The questionnaire features questions on participant satisfaction, the perceived effectiveness of the program, and the clarity and ease of following instructions. It invites suggestions for improvement and assesses the overall impact of the intervention. Scores range from 1 to 5, with higher scores indicating better clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schrefl, MSc, Principal Investigator — University of Bern; Daniel Erlacher, PhD, Study Chair — University of Bern; Andrea Schaerli, PhD, Study Chair — University of Bern; Nico Kolokythas, PhD, Study Chair — Elmhurst Ballet School
Locations (1):
- Elmhurst Ballet School, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Sensitive data of the students and the school.

REFERENCES:
- [Background] Goldmann JP, Bruggemann GP. The potential of human toe flexor muscles to produce force. J Anat. 2012 Aug;221(2):187-94. doi: 10.1111/j.1469-7580.2012.01524.x. PMID 22747582
- [Background] Goldmann JP, Sanno M, Willwacher S, Heinrich K, Bruggemann GP. The potential of toe flexor muscles to enhance performance. J Sports Sci. 2013;31(4):424-33. doi: 10.1080/02640414.2012.736627. Epub 2012 Oct 30. PMID 23106289
- [Background] Chiu LZF, Daehlin TE. Midfoot and Ankle Mechanics in Block and Incline Heel Raise Exercises. J Strength Cond Res. 2021 Dec 1;35(12):3308-3314. doi: 10.1519/JSC.0000000000004145. PMID 34570059
- [Background] Jarvis DN, Kulig K. Kinematic and kinetic analyses of the toes in dance movements. J Sports Sci. 2016 Sep;34(17):1612-8. doi: 10.1080/02640414.2015.1126672. Epub 2015 Dec 21. PMID 26691227
- [Background] Smith R, Lichtwark G, Farris D, Kelly L. Examining the intrinsic foot muscles' capacity to modulate plantar flexor gearing and ankle joint contributions to propulsion in vertical jumping. J Sport Health Sci. 2023 Sep;12(5):639-647. doi: 10.1016/j.jshs.2022.07.002. Epub 2022 Jul 21. PMID 35872091
- [Background] Tourillon R, Gojanovic B, Fourchet F. How to Evaluate and Improve Foot Strength in Athletes: An Update. Front Sports Act Living. 2019 Oct 11;1:46. doi: 10.3389/fspor.2019.00046. eCollection 2019. PMID 33344969
- [Background] Willemse L, Wouters EJM, Pisters MF, Vanwanseele B. Plantar intrinsic foot muscle activation during functional exercises compared to isolated foot exercises in younger adults. Physiother Theory Pract. 2024 Aug;40(8):1656-1668. doi: 10.1080/09593985.2023.2204947. Epub 2023 Apr 26. PMID 37126537